CLINICAL TRIAL: NCT06881030
Title: Comparison of the Efficacy of Different Modes of Accelerated Transcranial Magnetic Stimulation in Treatment-resistant Depression
Brief Title: Comparison of Different Acceleration Modes of Transcranial Magnetic Stimulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: [2025C]IIT. No. 026
Record Dates: First submitted 2025-03-10; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Treatment Resistant Depression (TRD)
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HL intervention group (Active Comparator): The motor threshold of 100% intensity, a TBS stimulus train stimulation for 2 seconds, including 10 times of 3 intrapascicular stimulation at 50 Hz and interapascicular stimulation at 5HZ, intervals of 10s, 60 repetitions, that is, a total of 1800 pulses per treatment, 10 treatments per day, intervals of 50 min, a total of 18000 pulses/day, continuous stimulation for 5 days.
  Interventions: Procedure: Noninvasive transcranial magnetic stimulation was administered 10 times daily
- TT intervention group (Experimental): The motor threshold of 100% intensity, a TBS stimulus train for 2 seconds, including 10 times of 3 intrapascicular stimulation at 50 Hz and interapascicular stimulation at 5HZ, intervals of 10s, 60 repetitions, that is, a total of 1800 pulses per treatment, 6 treatments per day, 50 min apart, a total of 10800 pulses/day, continuous stimulation for 5 days.
  Interventions: Procedure: Noninvasive transcranial magnetic stimulation was administered six times daily
- sham group (Sham Comparator): The appearance of the sham stimulation coil was consistent with that of the real stimulation coil, which could simulate the touch and sound of the scalp caused by the real stimulation. The treatment frequency, location, intensity and time of the sham stimulation group were the same as those of the real stimulation group.
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Noninvasive transcranial magnetic stimulation was administered six times daily — The motor threshold of 100% intensity, a TBS stimulus train for 2 seconds, including 10 times of 3 intrapascicular stimulation at 50 Hz and interapascicular stimulation at 5HZ, intervals of 10s, 60 repetitions, that is, a total of 1800 pulses per treatment, 6 treatments per day, 50 min apart, a total of 10800 pulses/day, continuous stimulation for 5 days.
  Arms: TT intervention group
Procedure: Noninvasive transcranial magnetic stimulation was administered 10 times daily — The motor threshold of 100% intensity, a TBS stimulus train stimulation for 2 seconds, including 10 times of 3 intrapascicular stimulation at 50 Hz and interapascicular stimulation at 5HZ, intervals of 10s, 60 repetitions, that is, a total of 1800 pulses per treatment, 10 treatments per day, intervals of 50 min, a total of 18000 pulses/day, continuous stimulation for 5 days.
  Arms: HL intervention group
Procedure: Sham — The appearance of the sham stimulation coil was consistent with that of the real stimulation coil, which could simulate the touch and sound of the scalp caused by the real stimulation. The treatment frequency, location, intensity and time of the sham stimulation group were the same as those of the real stimulation group.
  Arms: sham group

SUMMARY:
To compare the efficacy and safety of 6 times a day, 10 times a day acceleration mode and sham stimulation intervention for TRD, and to explore the antidepressant mechanism of accelerated mode, so as to provide a more simple and effective rapid treatment plan for TRD patients.

ELIGIBILITY:
Inclusion Criteria:

1. The current episode met the DSM-5 diagnostic criteria for major depression, without psychotic symptoms of the first or recurrent drug-free depressive subjects
2. After a full course of treatment with two or more antidepressants, the patient had no response, and the level of treatment resistance was moderate to severe as assessed by the Maudsley staging method

3.24-item Hamilton depression Scale score ≥20

4.The age ranged from 18 to 45 years, both sexes

5.Right handed

6.Written informed consent was obtained and patients volunteered to participate in the study and be evaluated.

Exclusion Criteria:

* 1. Comorbidity with other mental disorders, including schizophrenia, mental retardation, substance dependence, etc.

  2. Suffering from serious or unstable physical diseases

  3, pregnant, lactating women, women of childbearing age screening period urine HCG test results are positive

  4. Subjects with metal objects in the body or other contraindications to MRI scanning

  5. There are other conditions considered by the investigator to be inappropriate for participation in the clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale (24-items) Total Score Change | Baseline to end of stimulation period, an average of 5 days
  The Hamilton Depression Scale (24-items), is a 24 item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. It's considered the gold standard for rating depression severity and used frequently in clinical trials. Higher HAM-D24 score indicates more severe depression, and each item yields a score of 0 to 4. Remission is defined as HAM-D24 ≤8. A reduction of 50% or more in total score from Baseline indicates clinical response.

SECONDARY OUTCOMES:
Change in the rate of Hamilton Anxiety Scale score | Time Frame: Baseline to end of stimulation period, an average of 5 days
  Hamilton Anxiety Scale is a 17 item diagnostic questionnaire used to measure the severity of anxiety episodes in patients. Each item on the scale is rated on a 5-point scale from 0 (not present) to 4 (severe), with the total score ranging from 0 to 68. The HAMA-17 is often used in clinical and research settings to assess the severity of anxiety symptoms and to evaluate the effectiveness of treatments for anxiety. It is a more comprehensive version of the HAMA that includes additional items to capture a broader range of anxiety symptoms.

OTHER OUTCOMES:
Change in the rate of Beck Scale of Suicidal Ideation score | Baseline to end of stimulation period, an average of 5 days
  Beck Scale of Suicidal Ideation is a 21-item self-report instrument that detects and measures the intensity of a patient's specific attitudes, behaviors, and suicide plans during the past week. The BSI score ranges from 0 to 63, with higher scores indicating worse outcomes and lower scores indicating better outcomes.
Change in neuroimaging using functional magnetic resonance | Baseline to end of stimulation period, an average of 5 days
  Scanning functional magnetic resonance. Functional magnetic resonance imaging (fMRI) is a neuroimaging technique that is used to measure changes in brain activity by detecting changes in blood flow. In the context of major depression, fMRI has been used to study changes in brain function that may be associated with the condition. Research using fMRI in major depression has shown that there are alterations in the activity of certain brain regions in people with the condition.
Change in electroencephalogram | Baseline to end of stimulation period, an average of 5 days
  Electroencephalogram is collected from 64 electrodes. EEG can be used to identify patterns of brain activity that are associated with the condition and to inform treatment decisions. EEG can be a useful tool for identifying patterns of brain activity that are associated with TRD and for guiding treatment decisions. Neurofeedback and TMS are two approaches that have shown promise in the treatment of TRD. several parameters are analyzed to identify patterns of brain activity that may be associated with the condition. These parameters include:Alpha power, Beta power, Theta power, Delta power,etc.
Change of blood factor levels | Baseline to end of stimulation period, an average of 5 days
  Factors carried by peripheral blood and exosomes(Hypocretin, Brain-derived neurotrophic fact, Reelin, and N-methyl-D-aspartic acid receptor).

IPD SHARING:
Plan to Share IPD: Undecided